CLINICAL TRIAL: NCT04209530
Title: A Phase 2a, Open Label Study to Assess the Impact of CCH Treatment of Buttock and Thigh Cellulite in Adult Females Using Photonumeric Scales, Magnetic Resonance Imaging and Histopathology
Brief Title: Impact of CCH Treatment of Buttock and Thigh Cellulite in Adult Women
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to COVID-19 impact
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN3835-212
Record Dates: First submitted 2019-12-11; First posted 2019-12-24 (Actual); Results first posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2020-11

CONDITIONS: Cellulite; Edematous Fibrosclerotic Panniculopathy (EFP)
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Buttock & Posterolateral Thigh (Experimental): EN3835 up to 1.68 mg (Collagenase Clostridium Histolyticum)
  Interventions: Drug: EN3835

INTERVENTIONS:
Drug: EN3835 — Collagenase Clostridium Histolyticum (CCH)

SUMMARY:
This is a single center, open-label, Phase 2a study to assess the photonumeric scale, morphological, and histopathological changes associated with Collagenase Clostridium Histolyticum (CCH) in adult women with moderate or severe Edematous Fibrosclerotic Panniculopathy (EFP).

ELIGIBILITY:
Inclusion Criteria:

1. Have both buttocks or both posterolateral thighs with:

   1. A score of 3 or 4 (moderate or severe) as reported by the investigator using the Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS).
   2. A Hexsel Cellulite Severity Scale (CSS) Subsection A "Number of Evident Depressions" score of >0, and Subsection B "Depth of Depressions" score of 2 )medium depth depression) or 3 (deep depressions)..
2. Have a minimum of 2 well defined and isolated cellulite dimples.
3. Be willing to apply sunscreen to the treatment area before each exposure to the sun for the duration of the study (from the Screening Visit through the Day 251/Early Termination Visit).
4. Be judged to be in good health.
5. Have a negative pregnancy test.
6. Be willing and able to cooperate with the requirements of the study.

Exclusion Criteria:

1. Is from a vulnerable population, as defined by the United States (US) Code of Federal Regulations (CFR) Title 45, Part 46, Section 46.111(b) and other local and national regulations, including but not limited to, employees (temporary, part-time, full time, etc) or a family member of the research staff conducting the study, or of the sponsor, or of the contract research organization, or of the Institutional Review Board (IRB)/Independent Ethics Committee (IEC).
2. Has a history of sensitivity or allergy to collagenase or any other excipient of CCH.
3. Has systemic conditions (coagulation disorders, malignancy, keloidal scar, abnormal wound healing) that restricts study participation.
4. Has local (in areas to be treated) conditions (thrombosis, vascular disorder, active infection/inflammation, active cutaneous alteration, tattoo/mole) that restricts study participation.
5. Has skin laxity or linear undulations on the treatment region (both buttocks or both thighs) that can be effaced by lifting skin.
6. Requires anticoagulant or antiplatelet medication during the study.
7. Has used or intends to use any of the local applications/therapies/injections/procedures that restricts study participation.
8. Has used any form of artificial tanning (sprays, lotions, tanning booth, etc) within the 30 days prior to the first dose of study treatment or plans to use any form of artificial tanning during the study (through the Day 251/Early Termination Visit).
9. Has a positive HIV test and/or a positive Hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb) test at screening.
10. Has had any surgery, invasive procedure (eg, liposuction), injectable treatment (eg, KYBELLA®) or any similar treatment.
11. Has a history of keloids, hypertrophied scars, and/or other complications following biopsy.
12. Has any contraindications for MRI(implant containing metal, internal metallic object, permanent cosmetics/make-up, claustrophobia, syncope, low blood pressure, epilepsy, asthma, sickle cell disease) that restricts study participation.
13. Has received any collagenase treatments at any time prior to treatment in this study and/or has received EN3835 or CCH in a previous investigational study for cellulite.
14. Has previously received treatment with CCH in this clinical study.
15. Has received treatment with an investigational product within 30 days (or 5 half-lives, whichever is longer) of the Screening Visit.
16. Is pregnant and/or is providing breast milk or plans to become pregnant and/or to provide breast milk during the course of the study.
17. Has any other condition(s) that, in the investigator's opinion, might indicate the subject to be unsuitable for the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 7 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Dayoub, Study Director — Endo Pharmaceuticals
Locations (1):
- Endo Clinical Trial Site #1, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

RESULTS

PARTICIPANT FLOW:
Groups:
- Buttock; Posterolateral Thigh: EN3835 up to 1.68 mg (Collagenase Clostridium Histolyticum)
  EN3835: Collagenase Clostridium Histolyticum (CCH)
Period: Overall Study
Arm/Group | Buttock | Posterolateral Thigh
Started | 4 | 3
Completed | 0 | 0
Not Completed | 4 | 3
Not completed — Terminated due to the major disruption in study visits and protocol assessments due to COVID-19 | 4 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buttock | Posterolateral Thigh | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (5.46) | 38.3 (1.96) | 43.0 (5.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Skin Category (Fitzpatrick Scale) [Count of Participants; unit: Participants]
  I (Pale white) | 0 | 0 | 0
  II (Fair) | 0 | 0 | 0
  III (Darker white) | 1 | 1 | 2
  IV (Light brown) | 3 | 2 | 5
  V (Brown) | 0 | 0 | 0
  VI (Dark brown or black) | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: Kg] | 74.67 (12.836) | 78.32 (1.836) | 76.24 (9.344)
Height [Mean (Standard Deviation); unit: cm] | 163.83 (9.390) | 163.41 (2.933) | 163.65 (6.856)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.73 (1.744) | 29.50 (0.300) | 28.49 (1.566)

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline (Screening) in PR-PCSS
Description: Patient-Reported Photonumeric Cellulite Severity Scale (PR-PCSS) is a 5-point photonumeric scale rating cellulite severity from "0" (None) to "4" (Severe) from a patient's perspective
Time Frame: Day 71
Population: Because of the disruption of study conduct due to COVID-19, the study was prematurely terminated. No subjects completed assessments required for the Day 71 Visit and beyond. Only safety analyses were conducted.
Arm/Group | Buttock | Posterolateral Thigh
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: The Change From Baseline (Screening) in CR-PCSS
Description: Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS) is a 5-point photonumeric scale rating cellulite severity from "0" (None) to "4" (Severe) from a clinician's perspective
Time Frame: Day 22, Day 43 and Day 71
Population: as for outcome 1
Arm/Group | Buttock | Posterolateral Thigh
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: The Change From Baseline (Screening) in Hexsel Cellulite Severity Scale (CSS)
Description: Hexsel CSS is a photonumeric scale that looks at 5 key morphologic features of cellulite, each feature is evaluated on a 4-point scale from "0" (Low) to "3" (High)
Time Frame: Day 22, Day 43 and Day 71
Population: as for outcome 1
Arm/Group | Buttock | Posterolateral Thigh
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: MRI Before and After CCH Treatment
Description: Magnetic Resonance Imaging (MRI) of cellulite before and after CCH treatment
Time Frame: Day 71
Population: as for outcome 1
Arm/Group | Buttock | Posterolateral Thigh
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Histopathology Before and After CCH Treatment
Description: Histopathology of biopsies defined by the observation of the biopsied specimen by a trained Pathologist
Time Frame: Day 71
Population: as for outcome 1
Arm/Group | Buttock | Posterolateral Thigh
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All (Serious and Non-Serious AEs) from Day 1 to Day 265
Description: All serious and non-serious AEs, whether elicited or observed during study visit or spontaneously reported by the participant, including events that occurred from the time the participant signed the study specific consent form until completion of or discharge from the study.
Arm/Group | Buttock | Posterolateral Thigh
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Buttock (N=4) | Posterolateral Thigh (N=3)
Injection site bruising (General disorders) | 4 | 3
Injection site pain (General disorders) | 4 | 3
Injection site discolouration (General disorders) | 2 | 0
Injection site mass (General disorders) | 0 | 1
Injection site swelling (General disorders) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT04209530/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT04209530/SAP_001.pdf